CLINICAL TRIAL: NCT01980628
Title: A Multicenter, Open-Label, Phase 2 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor, Ibrutinib, in Subjects With Relapsed/Refractory Marginal Zone Lymphoma
Brief Title: Study of the Bruton's Tyrosine Kinase Inhibitor in Subjects With Relapsed/Refractory Marginal Zone Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1121-CA
Record Dates: First submitted 2013-10-29; First posted 2013-11-11 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Marginal Zone Lymphoma; B-cell Lymphoma
Keywords: MZL; NHL; SMZL; NMZL; MALT
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ibrutinib (Experimental): ibrutinib capsules: 560 mg once daily
  Interventions: Drug: ibrutinib

INTERVENTIONS:
Drug: ibrutinib
  Other Names: PCI-32765

SUMMARY:
Phase 2, open-label, non-randomized, monotherapy study to evaluate the safety and efficacy of ibrutinib in subject with relapsed/refractory Marginal Zone Lymphoma (MZL).

DETAILED DESCRIPTION:
Ibrutinib is a first-in-class, potent, orally administered covalent inhibitor of Bruton's tyrosine kinase (BTK). Inhibition of BTK blocks downstream B-cell receptor (BCR) signaling pathways and thus prevents B-cell proliferation. In vitro, ibrutinib inhibits purified BTK and selected members of the kinase family with 10-fold specificity compared with non-BTK kinases. Phase 1 and 2 studies of ibrutinib in B-cell malignancies demonstrate modest toxicity and significant single agent activity in a variety of B-cell malignancies, including NHL.

ELIGIBILITY:
Key Inclusion criteria:

* Histologically documented marginal zone lymphoma including splenic, nodal, and extranodal sub-types; subjects with splenic MZL must have an additional measurable lesion, nodal or extranodal, as described in inclusion criteria 5
* Previously received one or more lines of therapy including at least one CD20-directed regimen (either as monotherapy or as chemoimmunotherapy) with documented failure to achieve at least PR or documented PD after, the most recent systemic treatment regimen
* Men and women ≥18 years of age
* ECOG performance status of ≤2
* ≥1 measurable lesion site on CT scan (>1.5 cm in longest dimension). Lesions in anatomical locations (such as extremities or soft tissue lesions) that are not well visualized by CT may be measured by MRI instead. (Subjects with spleen-only disease are considered as not having measurable disease.)
* Life expectancy of >3 months, in the opinion of the investigator

Key Exclusion criteria:

* Medically apparent CNS lymphoma or leptomeningeal disease
* History of other malignancies except adequately treated non melanoma skin cancer, curatively treated in-situ cancer, or other solid tumors curatively treated with no evidence of disease for ≥2 years
* History of allogeneic stem-cell (or other organ) transplantation
* Any chemotherapy, anticancer antibodies, or other systemic anticancer therapy within 21 days of the first dose of study drug
* Any external beam radiation therapy within 6 weeks prior to the first dose of the study drug
* Concurrent use of warfarin or other vitamin K antagonists
* Concurrent use of a strong CYP3A inhibitor. Subjects who have received a strong CYP3A inhibitor prior to entering the study must have discontinued therapy for at least 5 half lives of the prohibited medication.
* Recent infection requiring IV anti-infective treatment that was completed ≤14 days before the first dose of study drug
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to CTCAE Grade 0 or 1, or to the levels dictated in the eligibility criteria with the exception of alopecia
* Inadequate organ function as defined on laboratory tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2017-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isaiah Dimery, MD, Study Director — Pharmacyclics LLC.
Locations (25):
- United States (13):
  - Site Reference ID/Investigator# 837, Tucson, Arizona
  - Site Reference ID/Investigator# 047, Duarte, California
  - Site Reference ID/Investigator# 377, Santa Monica, California
  - Site Reference ID/Investigator# 763, West Palm Beach, Florida
  - Site Reference ID/Investigator# 033, Atlanta, Georgia
  - Site Reference ID/Investigator# 370, Chicago, Illinois
  - Site Reference ID/Investigator# 195, Detroit, Michigan
  - Site Reference ID/Investigator# 350, New Hyde Park, New York
  - Site Reference ID/Investigator# 745, New York, New York
  - Site Reference ID/Investigator # 200, New York, New York
  - Site Reference ID/Investigator # 407, New York, New York
  - Site Reference ID/Investigator# 220, Hershey, Pennsylvania
  - Site Reference ID/Investigator# 348, Seattle, Washington
- Site Reference ID/Investigator# 560, Ghent, Oost-vlaanderen, Belgium
- France (7):
  - Site Reference ID/Investigator# 142, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Site Reference ID/Investigator# 737, Rouen, Haute-normandie
  - Site Reference ID/Investigator# 750, Lille, Hauts-de-France
  - Site Reference ID/Investigator# 749, La Roche-sur-Yon, Pays de la Loire Region
  - Site Reference ID/Investigator# 736, Nantes, Pays de la Loire Region
  - Site Reference ID/Investigator# 742, Rennes
  - Site Reference ID/Investigator# 735, Paris, Île-de-France Region
- Site Reference ID/Investigator# 669, Mainz, Rhineland-Palatinate, Germany
- United Kingdom (3):
  - Site Reference ID/Investigator# 030, Manchester, England
  - Site Reference ID/Investigator# 814, Oxford, England
  - Site Reference ID/Investigator# 368, Plymouth, England

REFERENCES:
- [Derived] Noy A, de Vos S, Coleman M, Martin P, Flowers CR, Thieblemont C, Morschhauser F, Collins GP, Ma S, Peles S, Smith SD, Barrientos JC, Chong E, Wu S, Cheung LW, Kwei K, Hauns B, Arango-Hisijara I, Chen R. Durable ibrutinib responses in relapsed/refractory marginal zone lymphoma: long-term follow-up and biomarker analysis. Blood Adv. 2020 Nov 24;4(22):5773-5784. doi: 10.1182/bloodadvances.2020003121. PMID 33227125
- [Derived] Noy A, de Vos S, Thieblemont C, Martin P, Flowers CR, Morschhauser F, Collins GP, Ma S, Coleman M, Peles S, Smith S, Barrientos JC, Smith A, Munneke B, Dimery I, Beaupre DM, Chen R. Targeting Bruton tyrosine kinase with ibrutinib in relapsed/refractory marginal zone lymphoma. Blood. 2017 Apr 20;129(16):2224-2232. doi: 10.1182/blood-2016-10-747345. Epub 2017 Feb 6. PMID 28167659

RESULTS

PARTICIPANT FLOW:
Groups:
- Ibrutinib: Subjects receive daily dose of 560 mg of ibrutinib capsules.
Period: Overall Study
Arm/Group | Ibrutinib
Started | 63 (Total number of patients enrolled to the study and received study treatment)
Completed | 0 (Participants who remain on treatment at Final Analysis.)
Not Completed | 63
Not completed — Adverse Event | 12
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 4
Not completed — PD, Subj non-Compliant,Study Terminated | 42

BASELINE CHARACTERISTICS:
Groups:
- Ibrutinib: Subjects receive a daily dose of 560 mg of ibrutinib capsules
Arm/Group | Ibrutinib
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants] — Participants were required to be of age 18 years or older
  Participants
    <=18 years | 0
    Between 18 and 65 years | 27
    >=65 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 53
  Black | 6
  Asian | 1
  Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: ORR (Overall Response Rate)
Description: ORR is defined as the proportion of subjects who achieved complete response (CR), partial response (PR). Response criteria are as outlined in the International Working Group Criteria for NHL, Cheson (2007), with disease assessments performed by an independent review committee (IRC).
  Per Cheson:
  CR is defined as disappearance of all evidence of disease. PR is defined as regression of measurable disease and no new sites.
Time Frame: Analysis was conducted with the cutoff date of 02 Nov 2017, with a median follow-up time of 33.1 months.
Measure: Mean (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Single Arm, Intent to Treat Population
Number analyzed (Participants) | 63
Percentage of Participants | 46 [33.5 to 59.3]

2. Secondary Outcome: DOR (Duration of Response)
Description: The DOR analyses is performed on the subset of subjects that achieve CR or PR as determined by IRC. DOR is calculated as the duration of time from the date of first response to the date of progression or death due to any cause.
Time Frame: Analysis was conducted with the cutoff date of 02 Nov 2017, with a median follow-up time of 33.1 months.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Ibrutinib: Patients receive daily dose of 560 mg of ibrutinib capsules.
Arm/Group | Ibrutinib
Number analyzed (Participants) | 63
Months | NA [16.7 to NA] — Per IRC assessment, the median DOR was not reached

ADVERSE EVENTS:
Time Frame: From the time of first ibrutinib dose until 30 days following the last dose of study drug
Description: For "At Risk" we considered 60 because it was the efficacy population (with N=60) is used for OS
Arm/Group | Ibrutinib
All-Cause Mortality (participants affected / at risk) | 17/63
Serious Adverse Events (participants affected / at risk) | 29/63
Other Adverse Events (participants affected / at risk) | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib (N=63)
Autoimmune Haemolytic Anaemia (Blood and lymphatic system disorders) | 2
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Pericardial Effusion (Cardiac disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 5
Cellulitis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Escherichia Sepsis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Listeria Sepsis (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Parainfluenzae Virus Infection (Infections and infestations) | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Fluid Overload (Metabolism and nutrition disorders) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Marginal Zone Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral Haemorrhage (Nervous system disorders) | 1
Cervical Radiculopathy (Nervous system disorders) | 1
Transient Ischaemic Attack (Nervous system disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Eosinophilic Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Bronchial Injury (Injury, poisoning and procedural complications) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib (N=63)
Anaemia (Blood and lymphatic system disorders) | 23
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Increased Tendency To Bruise (Blood and lymphatic system disorders) | 12
Atrial Fibrillation (Cardiac disorders) | 5
Vision Blurred (Eye disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 30
Nausea (Gastrointestinal disorders) | 20
Dyspepsia (Gastrointestinal disorders) | 12
Abdominal Pain (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 7
Abdominal Discomfort (Gastrointestinal disorders) | 4
Abdominal Distension (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 29
Oedema Peripheral (General disorders) | 15
Pyrexia (General disorders) | 12
Asthenia (General disorders) | 6
Upper Respiratory Tract Infection (Infections and infestations) | 16
Sinusitis (Infections and infestations) | 13
Bronchitis (Infections and infestations) | 7
Urinary Tract Infection (Infections and infestations) | 9
Oral Herpes (Infections and infestations) | 5
Conjunctivitis (Infections and infestations) | 4
Cystitis (Infections and infestations) | 4
Fall (Injury, poisoning and procedural complications) | 10
Contusion (Injury, poisoning and procedural complications) | 7
Skin Abrasion (Injury, poisoning and procedural complications) | 6
Weight Decreased (Investigations) | 9
Blood Alkaline Phosphatase Increased (Investigations) | 5
Blood Creatinine Increased (Investigations) | 4
Decreased Appetite (Metabolism and nutrition disorders) | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 10
Hyperuricaemia (Metabolism and nutrition disorders) | 10
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11
Hypokalaemia (Metabolism and nutrition disorders) | 9
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Hyponatraemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 13
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 10
Back Pain (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 14
Headache (Nervous system disorders) | 13
Anxiety (Psychiatric disorders) | 11
Depression (Psychiatric disorders) | 4
Haematuria (Renal and urinary disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 9
Ecchymosis (Skin and subcutaneous tissue disorders) | 6
Night Sweats (Skin and subcutaneous tissue disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 4
Rash Erythematous (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 10
Dry Eye (Eye disorders) | 4
Pain (General disorders) | 4
Cellulitis (Infections and infestations) | 7
Pneumonia (Infections and infestations) | 6
Ear Infection (Infections and infestations) | 4
Viral Upper Respiratory tract (Infections and infestations) | 4
Dehydration (Metabolism and nutrition disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Joint Swelling (Musculoskeletal and connective tissue disorders) | 4
Dysuria (Renal and urinary disorders) | 4
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Petechiae (Skin and subcutaneous tissue disorders) | 4
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement restrictions can vary and typically include (but are not limited to):

Required submission of all material for sponsor review at least thirty days prior to the proposed date of any presentation or submission. Materials must remove Proprietary Information, excluding Data /Study results. All Sponsor's comments are required to be included. Sponsor may delay the presentation/submission upon Sponsor review of materials that are being proposed for presentation/submission.